CLINICAL TRIAL: NCT04406818
Title: The Role of Metabolic and Hemodynamic Reserve in Age-Related Brain Vulnerability in Pediatric Sickle Cell Anemia
Brief Title: Metabolic and Hemodynamic Reserve in Pediatric SCA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 202106016; R01NS121065 (NIH)
Record Dates: First submitted 2020-05-22; First posted 2020-05-28 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Child, Only; Brain Diseases; Sickle Cell Disease; Anemia, Sickle Cell
Keywords: sickle cell anemia; cerebrovascular reactivity; cerebral oxygen metabolism; cortical thickness; gray matter; carbon dioxide; magnetic resonance imaging; brain development
MeSH Terms: conditions — Brain Diseases; Anemia, Sickle Cell | interventions — Carbon Dioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy Control (Active Comparator)
  Interventions: Drug: Carbon Dioxide
- Sickle Cell Anemia (Active Comparator)
  Interventions: Drug: Carbon Dioxide

INTERVENTIONS:
Drug: Carbon Dioxide — Participants inhale carbon dioxide while in magnetic resonance imaging scan to measure cerebrovascular reactivity

SUMMARY:
The purpose of this research study is to better understand how blood flow and metabolism change can influence brain development in the early decades of life. SCA participants and healthy controls are age and sex-matched for comparison. Within the SCA cohort, children with infarcts may have thinner cortices than those without, reflecting a greater loss.

The investigators will examine brain blood flow and metabolism using magnetic resonance imaging (MRI). The brain's blood vessels expand and constrict to regulate blood flow based on the brain's needs. The amount of expanding and contracting the blood vessels may vary by age. The brain's blood flow changes in small ways during everyday activities, such exercise, deep concentration, or normal brain growth. Significant illness or psychological stress may increase the brain's metabolic demand or cause other bigger changes in blood flow. If blood vessels are not able to expand to give more blood flow when metabolic demand is high, the brain may not get all of the oxygen it needs. In extreme circumstances, if the brain is unable to get enough oxygen for a long time, a stroke may occur. Sometimes small strokes occur without other noticeable changes and are only detectable on an MRI. These are sometimes called "silent strokes." In less extreme circumstances, not having a full oxygen supply may cause the brain to grow and develop more slowly than when it has a full supply.

One way to test the ability of blood vessels to expand is by measuring blood flow while breathing in carbon dioxide. Carbon dioxide causes blood vessels in the brain to dilate without increasing brain metabolism.

During this study participants may be asked to undergo a blood draw, MRI, cognitive assessments, and brief questionnaires. The study team will use a special mask to control the amount of carbon dioxide the participants breathe in.

ELIGIBILITY:
Healthy Controls:

* Healthy controls ages 4-21 years of age
* Able to participate in MRI scan without sedation
* Not currently pregnant
* No significant psychiatric history, defined as having a severe psychiatric diagnosis, per PI discretion
* No history of epilepsy
* No history of stroke or cerebrovascular disease
* May have occasional headaches if not taking a daily preventative medication for headaches
* Not on vasodilatory medication, such as sildenafil or verapamil

Sickle Cell Anemia Participants:

* Ages 4-21 years of age
* Hb SS or SBeta-thal
* Able to participate in MRI scan without sedation
* Not currently pregnant
* Not on vasodilatory medication, such as sildenafil or verapamil
* No known vasculopathy

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Gray Matter cortical thickness | 3 years
  Mean whole brain cortical thickness on high resolution T1 images

SECONDARY OUTCOMES:
Total Brain volume | 3 years
  Total brain volume (gray matter and white matter) on high resolution T1 image
Cerebrovascular Reactivity | 15 minutes
  Change in blood flow as measured by MRI in response to carbon dioxide

CONTACTS AND LOCATIONS:
Overall Officials: Kristin P Guilliams, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
The proposed research assets will include MRI scan data and CO2 breathing data from 120 subjects, including pediatric subjects. As children are a vulnerable population, the project team will make the data (with any personally identifiable information redacted) available to qualified investigators under a data sharing agreement that provides for (1) a commitment to using for research purposes only, (2) a commitment to securing the data using appropriate computer technology, and (3) a commitment to destroying the data after analyses are completed. This will be available upon request within 6 months of the grant period ending.
Supporting Information: ICF
Time Frame: At study conclusion
Access Criteria: Upon request by qualified researchers